CLINICAL TRIAL: NCT06748456
Title: Development and Evaluation of a Cluster Package Intervention to Promote an Evidence-based Use of PSA-tests in General Practice: A Cluster Randomized Trial
Brief Title: A Cluster Package Intervention to Promote an Evidence-based Use of PSA-tests in General Practice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Kvalitet i Almen Praksis (KiAP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 103342
Record Dates: First submitted 2024-10-16; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Evidence Based Medicine; Prostate Specific Antigen
Keywords: PSA-test; Prostate Cancer; Evidence based medicine; Quality clusters; General practice
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The study design is a cluster randomized trial. The quality clusters are the participants (clusters) and randomization will take place at quality cluster level. Each cluster includes on average 13 GP clinics.
  The control group will be offered the intervention at the end of the intervention period.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it will not be possible to blind the GP's or members of the research team after the allocation. The primary outcome is blinded to the statistician and data manager is blinded until outcomes are analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cluster package intervention group (Experimental): The intervention consists of:
  * A pre-recorded podcast to be heard by the GP's prior to the cluster meeting.
  * A two-hour meeting with a specific slideshow about PSA, data from the clinics within the cluster, current guidelines, cases and group discussions.
  * Two sets of hand-outs for the GP's to use in their own clinics.
  The intervention group will be offered the intervention during the intervention period of six months.
  Interventions: Behavioral: Podcast; Behavioral: Cluster meeting; Behavioral: Hand-out material 1; Behavioral: Hand-out material 2
- Standard care control group (No Intervention): The control group will be offered the intervention at the end of the intervention period.

INTERVENTIONS:
Behavioral: Podcast — A pre-recorded podcast with a urologist and a GP discussing the theme to promote preparatory reflections among the GPs before the cluster meeting
  Arms: Cluster package intervention group
Behavioral: Cluster meeting — A two-hour meeting facilitated by either the GPs cluster coordinator, another GP from the cluster or a facilitator outside the cluster chosen by the cluster itself with specific slides about PSA in general, guidelines, expert videos, data from the clinics, cases, and group discussions
  Arms: Cluster package intervention group
Behavioral: Hand-out material 1 — Hand-outs of the main take-home messages to facilitate further discussion in their respective GP offices
  Arms: Cluster package intervention group
Behavioral: Hand-out material 2 — Hand-outs to be used by GP and patients to facilitate communication about the relevance of taking a PSA-test
  Arms: Cluster package intervention group

SUMMARY:
It is widely acknowledged that prostate specific antigen (PSA) testing can lead to false-positives, overdiagnosis and overtreatment of prostate cancer. The current national clinical guidelines only recommend the test to a small group of patients and does not recommend neither systematic nor opportunistic screening for prostate cancer with the test.

The aim of this cluster randomized trial is to evaluate the effectiveness of a complex intervention aimed at improving the use of evidence based practice when using prostate specific antigen tests in general practice.

The complex intervention in this study is a so called cluster package which is meeting material to a quality cluster meeting as almost every general practitioner is a member of a quality cluster. Therefore, the investigators have developed a cluster package aimed at promoting an evidence-based use of the prostate specific antigen test to general practitioners.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most common type of cancer among men in Denmark with an incidence of approximately 4.500 cases and 1.300 deaths every year. Usually prostate cancer develops very slowly and men with a detectable prostate tumor can live for many years without experiencing any symptoms. Autopsy studies of males who died of other causes finds PC in approximately 30 percent of males in their fifties and up to 70 percent of males in their seventies. From that perspective most men die with prostate cancer than because of it.

In Denmark the first examinations of a possible prostate cancer diagnosis take place in general practice. Every citizen in Denmark with a social security number has free and direct access to a general practitioner (GP) and works as a gatekeeper to the healthcare system. If the GP suspects prostate cancer in a patient the GP has the possibility to measure the level of prostate specific antigen (PSA) in a blood sample. If the level of PSA is high it may indicate the presence of prostate cancer.

However, according to the national clinical guidelines on detection and diagnostic investigation of prostate cancer the PSA-test is only recommended on a small patient group with very specific and rare symptoms. Furthermore they do not recommend neither systematic nor opportunistic screening with the PSA-test.

The reason for the rather restrictive guidelines for PSA-testing is to avoid overdiagnosis and overtreatment of prostate cancer. A high level of PSA in a blood sample is not necessarily due to prostate cancer but could also be elevated by other conditions such as cystitis or an enlarged benign prostate. Even if the further examinations at a urology department in a hospital finds prostate cancer in the patient it is potentially indolent cancer and not a clinically important tumor which is an prostate cancer overdiagnosis and could lead to unnecessary treatment which is overtreatment. The treatment of prostate cancer could cause harms such as impotence, incontinence and faecal incontinence.

Since 2018, GP's in Denmark has been encouraged to cluster in groups of other GP's from their local area to work with quality development and form so called quality clusters. The aim of these quality clusters was to create a medical professional forum where the GP's could meet 2-4 times a year and exchange experiences with each other in a specific clinically relevant area decided by the cluster itself. One of the main points of the quality cluster concept was that the quality development work should be based on descriptive data from their own GP clinics. At present 116 quality clusters exist in Denmark and includes 3.519 GP's in 1.542 GP clinics.

By the same time of the establishment of the quality cluster a national organization called KiAP (a Danish acronym for Quality in General Practice) was founded. The primary purpose was to support the quality clusters with their quality development work. One of the supportive initiatives by KiAP is the development of cluster packages which is meeting material for the quality clusters on their cluster meetings. A cluster packages has one specific clinically relevant theme and consists of data, expert videos, reflection questions among other things.

The investigators have chosen to develop a cluster package about PSA-tests in general practice with the purpose to promote an evidence-based practice. A pilot study will be conducted in the development process. The aim of the study is to evaluate the effectiveness of the cluster package. Since the study is a cluster randomized trial the investigators invited all the Danish quality clusters to agree to use the cluster package on one of their cluster meetings. The participating quality clusters are randomized to an intervention group and a control group.

ELIGIBILITY:
Inclusion Criteria:

* Quality clusters with a cluster coordinator
* Quality clusters willing to participate in a cluster meeting with PSA as a theme in 2025.

Exclusion Criteria:

* Quality clusters who already planned their cluster meetings in 2025.
* Quality clusters unwilling to await allocation before planning their cluster meetings in 2025.
* Quality clusters participating in the pilot study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change of prostate specific antigen tests on unique men ≥40 taken by general practitioners | From cluster meeting to the end of intervention period at 6 months
  The primary outcome is a reduction in the prevalence of prostate specific antigen (PSA) test on unique men ≥40 taken at the level of the quality health cluster from six month pre-intervention until six months post-intervention, in the intervention group compared to the control group. The overall aim is to improve practice of evidence based medicine by general practitioners (GP's), therefore we do not attempt to remove all PSA-test taken, neither do we set a pre-defined number that needs to be achieved. However, when following Danish Guidelines for PSA-testing, only a very small proportion of males over 40 should have the test, and therefore we consider any reduction clinically relevant.

SECONDARY OUTCOMES:
Pre/post intervention change | From cluster meeting to the end of intervention period at 6 months
  The prevalence of PSA test on unique men ≥40 taken at each GP clinic from pre- to post-intervention
High-user change | From cluster meeting to the end of intervention period at 6 months
  The change in the prevalence of PSA test on unique men ≥40 taken by the 10% highest users defined as all GP clinics
Variance between GPs | From cluster meeting to the end of intervention period at 6 months
  The homogeneity in the prevalence of PSA tests on unique men ≥40 within each cluster in the intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Marius Brostrøm Kousgaard, Associate professor, Principal Investigator — Center of General Practice, Department of Public Health, University of Copenhagen
Locations (1):
- Center of General Practice, Department of Public Health, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No